CLINICAL TRIAL: NCT05333809
Title: Explore the Efficacy and Safety of Pembrolizumab and Disitamab Vedotin in HER2 Expressing Metastatic Colorectal Cancer Failed at Least Two Lines of Systemic Treatment
Brief Title: Pembrolizumab and Disitamab Vedotin in HER2-expressing Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Director of Oncology Department, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HERPANDA
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pembrolizumab; disitamab vedotin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Pembrolizumab plus Disitamab vedotin
  Interventions: Drug: Pembrolizumab; Drug: Disitamab vedotin

INTERVENTIONS:
Drug: Pembrolizumab — an anti-PD-1 monoclonal antibody
Drug: Disitamab vedotin — HER2-ADC

SUMMARY:
This is an open-label, multi-center, phase Ⅱ study. This study will evaluate the efficacy and safety of pembrolizumab in combination with disitamab vedotin in subject with HER2-expressing metastatic Colorectal Cancer (mCRC).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of histologically or cytologically confirmed unresectable metastatic CRC (KRAS, NRAS and BRAF wild type) with HER-2 expression (IHC2+ or IHC 3+) will be enrolled in this study.
2. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
3. Histologically and/or cytologically confirmed colorectal cancer, including:

   （a) Unresectable metastatic colorectal adenocarcinoma (b)Evaluable or measurable HER2 expressing (IHC 3+ or IHC 2+) disease
4. Have received at least 2 prior treatments with systemic chemotherapy regimen until disease progression or intolerance; the patients with disease progression during or within 6 months after the adjuvant or neoadjuvant chemotherapy treatment should be recorded as first-line treatment; There is no restriction on whether the patient has received previous anti-HER2 treatment; for patients who have received previous anti-HER2 treatment, tissue re-biopsy should be done to confirm the expression of HER2 before enrollment; for patients who haven't received previous anti-HER2 treatment, HER2 status may refer to previous testing results from Tier 1 hospital.
5. Have measurable disease based on RECIST 1.1.
6. Have life expectancy of at least 3 months
7. Have adequate organ function as defined in the following table (Table 4).
8. Male participants: A male participant must agree to use a contraception as detailed in Appendix 2 of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.
9. Female participants: The participant (or legally acceptable representative if applicable) provides written informed consent for the trial. A female participant is eligible to participate if she is not pregnant (see Appendix 2), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 2 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 2 during the treatment period and for at least
10. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.

Exclusion Criteria:

1. Patients with any previous histological or hematological test showing mismatch repair gene deletion (dMMR), microsatellite instability (MSI-H)
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-CTLA-4 or any cellular immunotherapy; has received prior therapy with other HER2-ADC tubulin inhibitors (such as T-DM1, RC-48, DS8201, etc.) or participated in similar clinical studies;
3. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
4. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
5. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease, pulmonary fibrosis, acute lung disease, or uncontrolled systemic diseases (i.e., diabetes, hypertension).
6. Clinically uncontrollable diarrhea
7. Has a chronic or active infection requiring systemic antibacterial, antifungal, or antiviral therapy, including tuberculosis infection, etc. Patients with a history of active TB infection ≥1 year prior to screening should also be excluded, unless proof can be provided that appropriate treatment has been completed.
8. Has known active CNS metastases and/or carcinomatous meningitis.
9. Clinically significant pleural effusion, pericardial effusion or ascites requiring multiple drains within 2 weeks prior to treatment
10. Known second primary malignancy or additional malignancy within the past 5 years (Participants with basal cell carcinoma of the skin or carcinoma in situ of the cervix that have undergone potentially curative therapy are not excluded)
11. Uncontrolled diabetes or electrolyte disorder after the standard medical treatment
12. Has a known history of Human Immunodeficiency Virus (HIV) infection.
13. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection. Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA > 500 IU/mL and patients with positive HCV) RNA should be excluded.

    Note: Hepatitis B and C screening tests are not required unless:
    * Known history of HBV and HCV infection
    * As mandated by local health authority
14. Has any major surgery≤28 days prior to the first dose
15. Prior allogeneic stem cell transplantation or prior organ transplantation.
16. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and RC48-ADC and/or any of its excipients.
17. History of duodenal ulcer, ulcerative colitis, intestinal obstruction, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers; history of intestinal perforation and fistula, but have not recovered after surgical treatment.
18. History of arterial thrombosis or deep vein thrombosis within 6 months before enrollment, or evidence or history of bleeding tendency within 2 months before enrollment, regardless of severity
19. History of Stroke or transient ischemic attack occurred within the first 12 months prior to enrollment.
20. Severe ulcer or fracture of skin, surgical site, wound site and mucosa is not completely healed.
21. Acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting ≤ 6 months prior to study enrolment; New York Heart Association (NYHA) Functional Classification Grade II or greater congestive heart failure.
22. Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks, or immunotherapy (such as interleukin, interferon, thymosin), hormone therapy, targeted therapy or any research therapy within 14 days or 5 half-lives prior to start of study treatment [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to allocation.
23. Have received any Chinese herbal medicine or proprietary Chinese medicine for anticancer within 14 days prior to start of study treatment.
24. Patients whose toxic and side effects (due to previous anticancer treatment) have not recovered to baseline or stable level, unless AE may not with safety risks (such as hair loss, neuropathy and specific laboratory abnormalities).
25. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.
26. Has an active or chronic infection requiring systemic therapy including tuberculosis infection, etc. History of active tuberculosis infection ≥1 year before screening should also be excluded, unless proof can be provided that appropriate treatment has been completed.

    Note: No HIV testing is required unless mandated by local health authority.
27. Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
28. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
29. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
30. Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months after the last subject participating in
  proportion of patients with complete and partial remission in the best efficacy

SECONDARY OUTCOMES:
Disease control rate (DCR) | 24 months after the last subject participating in
  the best efficacy is the proportion of patients with complete remission, partial remission and stable disease
Progression free survival time (PFS) | 24 months after the last subject participating in
  time from the start of medication to the initial progression of the disease
Overall survival (OS) | 36 months after the last subject participating in
  time from the start of medication to death

IPD SHARING:
Plan to Share IPD: Yes